CLINICAL TRIAL: NCT05048615
Title: Efficacy and Safety of Ambulatory Low-dose Venetoclax and Azacitidne as First Line Therapy in Newly Diagnosed AML: a Pilot Study
Brief Title: Low-dose Venetoclax and Azacitidine as Front-line Therapy in Newly Diagnosed AML
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, David Gomez Almaguer, Head of Hematology Service, Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE21-00014
Record Dates: First submitted 2021-07-26; First posted 2021-09-17 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: AML
Keywords: acute myeloid leukemia; venetoclax; azacitidine; first-line therapy; induction chemotherapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax; Itraconazole; Azacitidine

STUDY DESIGN:
Intervention Model Description: A consecutive sample of 15 patients with newly diagnosed AML will be prospectively included in this study.
Masking Description: This is an Open label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Low-dose Ventoclax and oral itraconazol plus subcutaneous Azacitdine (Experimental): Patients will recieve Low-dose Venetoclax at a dose of 100mg/day por 21 days, oral itraconazol 100mg every 12 hours, and subcutaneous Azacitidine 75mg/m2 (maximun dose 100mg) daily for seven days. Each cycle duration is 21 days and patients will recieve a maximun of two cycles.
  Interventions: Drug: Venetoclax 100 MG; Drug: Itraconazole capsule; Drug: Azacitidine Injection

INTERVENTIONS:
Drug: Venetoclax 100 MG — Patients will receive oral Venetoclax at a fixed dose of 100mg/day from day 1 to day 21 per cycle for a maximum of 2 cycles.
  Other Names: Venclexta
Drug: Itraconazole capsule — Patients will receive oral itraconazole at a dose of 100 mg every 12 hours from day 1 to day 21.
Drug: Azacitidine Injection — Patients will receive a maximum of two cycles of daily subcutaneous Azacitidine at a dose of 75 mg/m2 (maximum 100 mg) from day 1 to day 7.
  Other Names: Vidaza

SUMMARY:
Venetoclax plus azacitidine are effective in treating newly diagnosed AML in patients who cannot recieve intensive chemotherapy. However there is no clinical data rewarding the efficacy and safety of low-dose venetoclax and azacitidine as first-line therapy.

DETAILED DESCRIPTION:
Venetoclax plus azacitidine are effective in treating newly diagnosed AML in patients who cannot recieve intensive chemotherapy. However there is no clinical data rewarding the efficacy and safety of low-dose venetoclax and azacitidine as first-line therapy. This phase 2 clinical trial will explore the efficacy and safety of low-dose venetoclax (100mg /day/21 days) and a fixed dose of azacitidine (75mg/m2, maximun dose 100mg, SC for seven consecutive days) for a maximun of two cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. Both genders
3. Diagnosis of non-m3 AML by the WHO 2016 diagnostic criteria
4. Patients eligible and not eligible for transplant
5. AML secondary to treatment or associated to myelodisplasia

Exclusion Criteria:

1. AML with PML/RAR-alfa translocation t(15;17)
2. Central nervous system involvement
3. Poor functional status (ECOG>2)
4. Organic dysfunction (Marshall score ≥2)
5. Active infection
6. Use of other CYP3A4 inhibitors
7. Pregnancy
8. GFR <30 ml/min/1.72m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Feasibility will be address by obtaining the proportion of patients who need hospitalization | 1 month
  If therapy is feasible >50% of patients will recieve their first cycle of treatment without hospitalization
Safety will be defined by the number of patients deceased before 14 days of initiating treatment | 2 weeks
  If therapy is safe then <10% of patients will die in the first 14 days of treatment
Safety will be defined by the number of patients deceased before 30 days of initiating treatment | 1 month
  If therapy is safe then <20% of patients will die in the first 30 days of treatment

SECONDARY OUTCOMES:
Efficacy will be achieved if the overall response rate is similar to standard of care (7+3) | 2 months
  If the therapy is effective then overall response rates will be similar to those reported with standard of care (7+3)

CONTACTS AND LOCATIONS:
Overall Officials: David Gomez-Almaguer, Principal Investigator — Universidad Autonoma de Nuevo Leon
Locations (1):
- Andres Gomez, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dohner H, Weisdorf DJ, Bloomfield CD. Acute Myeloid Leukemia. N Engl J Med. 2015 Sep 17;373(12):1136-52. doi: 10.1056/NEJMra1406184. No abstract available. PMID 26376137
- [Background] Guerra VA, DiNardo C, Konopleva M. Venetoclax-based therapies for acute myeloid leukemia. Best Pract Res Clin Haematol. 2019 Jun;32(2):145-153. doi: 10.1016/j.beha.2019.05.008. Epub 2019 May 24. PMID 31203996
- [Background] Pollyea DA, Amaya M, Strati P, Konopleva MY. Venetoclax for AML: changing the treatment paradigm. Blood Adv. 2019 Dec 23;3(24):4326-4335. doi: 10.1182/bloodadvances.2019000937. PMID 31869416
- [Background] DiNardo CD, Pratz K, Pullarkat V, Jonas BA, Arellano M, Becker PS, Frankfurt O, Konopleva M, Wei AH, Kantarjian HM, Xu T, Hong WJ, Chyla B, Potluri J, Pollyea DA, Letai A. Venetoclax combined with decitabine or azacitidine in treatment-naive, elderly patients with acute myeloid leukemia. Blood. 2019 Jan 3;133(1):7-17. doi: 10.1182/blood-2018-08-868752. Epub 2018 Oct 25. PMID 30361262
- [Derived] De la Garza-Salazar F, Colunga-Pedraza PR, Gomez-Almaguer D, Garcia-Zarate VA, Gomez-De Leon A. Low dose venetoclax plus itraconazole outpatient induction in newly diagnosed acute myeloid leukemia: A phase 2 study. Leuk Res. 2023 Oct;133:107373. doi: 10.1016/j.leukres.2023.107373. Epub 2023 Aug 22. PMID 37633156